CLINICAL TRIAL: NCT06530420
Title: The Usefulness of the New EHS/AHS Classification of Primary Umbilical Hernias in the Selection of Method of Their Treatment
Status: Recruiting | Type: Observational
Sponsor: Brothers Hospitallers Hospital in Cracow (Other)
Responsible Party: Principal Investigator, Nicole Kantor, doctor, Brothers Hospitallers Hospital in Cracow
Other Study IDs: 118.0043.1.167.2024
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Retrospective Analysis of Material From the Hospital Database

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Umbilical hernia repair surgery — collected information about: gender, age, comorbidities, body weight, time of surgery, hernia size and treatment methods and reccurence

SUMMARY:
The aim of the study is to assess the usefulness of the new classification of primary umbilical hernias in the choice of treatment of patients.

The study is conducted as a retrospective analysis of material from the hospital database

DETAILED DESCRIPTION:
A retrospective analysis will include patients operated on in the Department of General Surgery of the Hospital of the Brothers Hospitallers in the period from January 2016 to December 2022. The incidence of recurrence will be assessed based on outpatient records and a telephone survey. Hernias will be classified according to the EHS/AHS guidelines as small, medium and large. The qualification will take into account the old and new classification of hernias.

ELIGIBILITY:
Inclusion Criteria:

* Repair surgery for primary umbilical hernia

Exclusion Criteria:

* Repair surgery for recurrent umbilical hernia

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with umbilical hernia operated in the Department of General Surgery of the Hospital of the Brothers Hospitallers in the period from January 2016 to December 2022
Sampling Method: Probability Sample
Enrollment: 1087 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of umbilical hernia recurrence | 20.12.2025

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the Brothers Hospitallers of Saint John of God, Krakow, Poland

REFERENCES:
- [Derived] Kantor N, Gach T, Orzeszko Z, Kaciczak M, Frycz J, Solecki R, Markowska B, Bogacki P, Szura M. The Usefulness of the New EHS/AHS Classification of Primary Umbilical Hernias in the Selection of the Method of Their Treatment. Pol Przegl Chir. 2025 Jul 29;97(5):25-30. doi: 10.5604/01.3001.0055.2300. PMID 41171115